CLINICAL TRIAL: NCT06684587
Title: Telehealth Exercise and Mindfulness for Pain in Osteoarthritis: A Stage 1B Feasibility Study
Brief Title: Telehealth Exercise and Mindfulness for Pain in Osteoarthritis - Stage 1B
Acronym: TEMPO-1B
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Deepak Kumar, Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7510
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis
Keywords: Telehealth; Exercise; Mindfulness; Pain; Feasibility
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity; Pain | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Parallel-arm randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TX (Telehealth Exercise) (Active Comparator): Participants in this group will receive a group-based, supervised exercise session twice a week for 10 weeks along with a structured home exercise program. These sessions will be delivered via Boston University HIPAA-compliant Zoom videoconferencing software.
  Interventions: Behavioral: Exercise Program
- Group TMX (Telehealth Exercise and Mindfulness) (Experimental): Participants in this group will receive a group-based, supervised, integrated mindfulness and exercise program twice a week for 10 weeks along with a structured home program. Similar to the exercise intervention, these sessions will be delivered via Boston University HIPAA-compliant Zoom videoconferencing software.
  Interventions: Behavioral: Mindful Exercise

INTERVENTIONS:
Behavioral: Exercise Program — In this 10-week intervention, participants will be given strengthening exercises and neuromuscular re-education exercises.
  Arms: Group TX (Telehealth Exercise)
Behavioral: Mindful Exercise — In this 10-week intervention, mindfulness meditation will be integrated with strengthening and neuromuscular exercises recommended for knee osteoarthritis.
  Arms: Group TMX (Telehealth Exercise and Mindfulness)

SUMMARY:
The goal of this randomized controlled trial (RCT) is to test the feasibility of an 10-week telehealth mindful exercise intervention compared to a telehealth exercise only intervention for people with knee osteoarthritis (OA). This RCT will be fully digital with all recruitment, assessments, and intervention being conducted remotely.

DETAILED DESCRIPTION:
In this RCT, 62 adults with knee osteoarthritis will be assigned to either an exercise arm or mindful exercise arm. Both interventions will be delivered via videoconferencing in a group setting. In both groups, participants will receive a supervised session twice a week for 10 weeks. Participants will also receive a home program. During the study period, participants will be asked to remotely complete brief surveys every week and longer surveys on pain, function, mood, and other symptoms at baseline, week 5, week 10, week 16, and week 22. These surveys will be about pain, function, mood, and other symptoms. Participants will complete digital wearable-sensor based assessments at baseline and week 10. Participants will also be asked to complete brief surveys each week during the study. Feasibility of the intervention will be determined post-intervention by outcome measures such as recruitment rate, retention rate, and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Meet National Institute for Health and Clinical Excellence clinical guidelines for knee osteoarthritis (i.e., age ≥ 50 years, presence of activity related pain, no morning knee stiffness or presence of morning knee stiffness ≤ 30 minutes)
* BMI<40
* Knee pain on most days for 3 months or more
* Average overall knee pain severity of ≥ 4 on an 11-point numeric rating scale over last 7 days, at least 2 weeks apart
* Able to attend remote sessions
* Can speak and understand English at a sufficient level to understand the study procedures and informed consent.
* Available for study duration

Exclusion Criteria:

* Contraindications to exercise
* Other pain in lower back or legs that is greater than knee pain
* Received physical therapy treatment for knee OA in the past 6 months or currently receiving physical therapy
* Received any mindfulness programs such as Tai Chi, meditation, etc. in the past 6 months or currently receiving such program
* Currently receiving chemotherapy or radiation therapy for cancer except non-melanoma skin cancer
* History of other disease that may involve the index joint including inflammatory joint disease such as rheumatoid arthritis, seronegative spondyloarthropathy (eg, ankylosing spondylitis, psoriatic arthritis, inflammatory bowel disease related arthropathy), crystalline disease (eg, gout or pseudogout), lupus erythematosus, knee joint infections, Paget's disease affecting the knee, or knee joint tumors.
* Any knee surgery in the previous 6 months
* Joint replacement in either hip or ankle
* Previous knee osteotomy partial or total knee replacement in either knee
* Planned major treatment for knee OA (e.g., surgery, injections, physical therapy) during the study period
* Planned major surgery in the next 6 months
* Corticosteroid or hyaluronic acid injections in either knee in the previous 3 months
* Neurological conditions that impacts motor functioning (e.g., stroke, Parkinson's disease, Alzheimer's disease, Multiple Sclerosis, diabetic neuropathy, etc).
* Pregnancy (self-report)
* Participation in another clinical trial for any joint or muscle pain
* Suspected or known drugs or alcohol abuse

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Throughout the recruitment process; up to 12 months from the start of the study
  Proportion of participants that are recruited for the study
Attendance | Throughout the intervention period (over 10-weeks)
  Proportion of sessions attended.
Retention Rate | Post-intervention visit (10-week)
  Proportion of participants who complete patient-reported outcome surveys.
Adverse and serious adverse events | From first intervention session to week 22
  # of intervention related adverse or serious adverse events

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | Baseline, 5-week, 10-week, 16-week, 22-week
  Patient-reported outcome for knee pain and disability; a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Numeric Rating Scale - Nominated Activity | Weekly for 22 weeks
  Average rating of knee pain from 0-10, where 0 represents no pain and 10 represents worst pain imaginable, in the past week in a nominated activity selected at baseline.
Participant Feedback Survey | 5-week, Post-intervention visit (10-week), Follow-up visit (22-week)
  Custom scale measuring feedback on interventionists and interventions. Scores range from 0-4 (0 - Strongly Disagree, 1 - Disagree, 2 - Neither Agree no Disagree, 3 - Agree, and 4 - Strongly Agree).
Satisfaction Scale | Post-intervention visit (10-week), Follow-up visit (22-week)
  Custom 4-item (0-10 Likert scale) to determine satisfaction with individual components of the intervention.
Pain Catastrophizing Scale | Baseline, 5-week, 10-week, 16-week, 22-week
  13-item self-report measure designed to assess catastrophic thinking related to pain among adults with or without chronic pain. Each item is rated on a 5-point scale: 0 (Not at all) to 4 (all the time).
Participant Global Impression of Change | 5-week, 10-week, 16-week, 22-week
  Participant's rating of change in condition on a 15-point scale. Higher scores represent improvement and lower scores represent worsening or no change in symptoms.
Tampa Scale of Kinesiophobia | Baseline, 10-week, 22-week
  17-item self-report checklist with a 4-point Likert scale (1 - Strongly disagree; 2 - Disagree; 3 - Agree; 4 - Strongly agree) to assess one's fear of movement. Scoring of items 4, 8, 12, and 16 must be reversed, where "strongly disagree" is 4 points, "disagree" is 3 points, "agree" is 2 points, and "strongly agree" is 1 point. Sum up the scores for all 17 items to obtain the total raw score, ranging from 17 to 68 points. Higher total scores indicate an increasing degree of kinesiophobia, with 17 indicating no kinesiophobia or negligible fear of movement and 68 representing the highest possible level of kinesiophobia.
Global Mindfulness Scale | Baseline, 10-week, 22-week
  13-item tool that assesses all five mindfulness factors: Allowance, Boundlessness, Open-Heartedness, Insight, and Presence.

OTHER OUTCOMES:
7-meter Walk Test | Baseline,10-week
  Functional test that measures comfortable walking speed as participant walks for two laps of a 7-meter path for a total walking distance of 28-meters. Participants will performance this visit remotely at their home.
Pain, Enjoyment, General Activity Scale | Baseline, 5-week, 10-week, 16-week, 22-week
  3-item scale assessing pain intensity and interference. The response range is 0-10; the score of Pain, Enjoyment, General Activity Scale is the mean of the three individual item scores. Higher scores represent worse pain and pain-related interference.
Patient Global Assessment of Osteoarthritis | Baseline, 5-week, 10-week, 16-week, 22-week
  Participant's assessment of impact of osteoarthritis on their general health on a 0-100 mm scale. Higher scores represent higher impact of disease or worse global health.
Treatment History | Baseline, 5-week, 10-week, 16-week, 22-week
  A survey that collects information about the treatments the individual has undertaken for their knee osteoarthritis
Widespread Pain Index Symptom Severity Scale | Baseline, 5-week, 10-week, 16-week, 22-week
  Self-reported outcome on severity of cognitive symptoms such as fatigue, trouble thinking or remembering, waking up tired, and other physical symptoms such as headache, dizziness, etc. Each symptom is scored on a 4-point scale where 0 indicates no problem and 3 indicates severe problem. Scores are calculated by summing items, with higher scores (out of a maximum score of 12) indicating greater symptom severity.
Generalized Anxiety Disorder 7-item | Baseline, 5-week, 10-week, 22-week
  7-item questionnaire for anxiety, with scoring from 0-3 on each item. A total score of 0-4 indicates minimal anxiety; 5-9 for mild anxiety; 10-14 for moderate anxiety; and 15-21 for severe anxiety
Patient Health Questionnaire 8-item | Baseline, 10-week, 22-week
  8-item scale assessing depression symptoms. Each question is scored from 0 to 3, where higher scores indicate higher frequency of experiencing depressive symptoms. The total score is the sum value of individual questions. Higher total scores indicate greater severity of depression.
Homunculus | Baseline, 5-week, 10-week, 16-week, 22-week
  Assess the number of painful, aching or stiffed joints.
Arthritis Self Efficacy Scale | Baseline, 10-week, 22-week
  Self-reported outcome assessing confidence in one's capacity to function despite pain. Scores range from 10 (very uncertain) to 100 (very certain). Higher scores indicate greater self-efficacy to manage osteoarthritis.
Fear Avoidance Beliefs Questionnaire - Physical Activity | Baseline,10-week
  Self-reported outcome assessing how one's fear avoidance beliefs contributes to the cognitive/affective part of their knee pain. Each item is scored from 0 to 6. Total scores are the summation of each item scores. Higher total scores indicate greater fear of physical activity.
Whole Person Health Index | Baseline,10-week
  9-question survey tool that integrates individual-level biological and behavioral factors
Daily life gait speed | Baseline,10-week
  Participants will be asked to wear a single inertial sensor that will be placed on their lower back for a period of 7 days. Mean daily walking in meters per second speed over 7 days will be extracted
Daily life gait speed variability | Baseline,10-week
  Participants will be asked to wear a single inertial sensor that will be placed on their lower back for a period of 7 days. Standard deviation of daily walking speed in meters per second over 7 days will be extracted
Weekly medication use | Weekly for 22-weeks
  # of days and # of times/day of analgesic medication use for knee pain
Weekly strengthening exercise | Weekly for 22-weeks
  # of minutes of strengthening exercise per day of the week
Weekly aerobic exercise | Weekly for 22-weeks
  # of minutes of aerobic exercise per day of the week
Weekly mindfulness practice (only for mindful exercise group) | Weekly for 22-weeks (only for mindful exercise group)
  # of minutes of mindfulness practice per day of the week

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Requests will be considered on an individual basis

REFERENCES:
- [Background] Shah N, Morone N, Kim E, Ellis TD, Cohn E, LaValley MP, Kumar D. Telehealth mindful exercise for people with knee osteoarthritis: A decentralized feasibility randomized controlled trial. Osteoarthr Cartil Open. 2024 Jun 19;6(3):100494. doi: 10.1016/j.ocarto.2024.100494. eCollection 2024 Sep. PMID 39021877